CLINICAL TRIAL: NCT06591104
Title: Metabolic Phenotypes of Obesity and Diabetic Kidney Disease in Patients with Type 2 Diabetes Mellitus
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, George Armia Ghaly Abdelmaseih, Resident physician at Internal Medicine department, Assiut University
Other Study IDs: obesity and DKD in T2DM
Record Dates: First submitted 2024-08-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Kidney Disease; Obesity; Metabolic Syndrome; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetic Nephropathies; Obesity; Metabolic Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- metabolically healthy non obesity (MHNO): According to the NCEP ATP III definition, metabolic syndrome is present if three or more of the following five criteria are met: waist circumference over 40 inches (men) or 35 inches (women), blood pressure over 130/85 mmHg, fasting triglyceride (TG) level over 150 mg/dl, fasting high-density lipoprotein (HDL) cholesterol level less than 40 mg/dl (men) or 50 mg/dl (women) and fasting blood sugar over 100 mg/dl.
  Obesity was defined as a BMI of ≥ 25.0 kg/m2 . Patients with a BMI of 18.5-<23.0 were considered normal weight; for those with a BMI of 23.0-<25.0 were overweight. The patients with normal weight and those who were overweight were collapsed into the non-obesity group.
  so this group of patients are metabolically healthy and non obese with BMI 18.5 - <25
  Interventions: Diagnostic Test: 24 hour urinary protein
- metabolically healthy obesity ( MHO ): According to the NCEP ATP III definition, metabolic syndrome is present if three or more of the following five criteria are met: waist circumference over 40 inches (men) or 35 inches (women), blood pressure over 130/85 mmHg, fasting triglyceride (TG) level over 150 mg/dl, fasting high-density lipoprotein (HDL) cholesterol level less than 40 mg/dl (men) or 50 mg/dl (women) and fasting blood sugar over 100 mg/dl.
  Obesity was defined as a BMI of ≥ 25.0 kg/m2 . Patients with a BMI of 18.5-<23.0 were considered normal weight; for those with a BMI of 23.0-<25.0 were overweight. The patients with normal weight and those who were overweight were collapsed into the non-obesity group.
  so this group of patients are metabolically healthy but they are obese with BMI of ≥ 25.0 kg/m2
  Interventions: Diagnostic Test: 24 hour urinary protein
- metabolically unhealthy non obsesity ( MUNO ): According to the NCEP ATP III definition, metabolic syndrome is present if three or more of the following five criteria are met: waist circumference over 40 inches (men) or 35 inches (women), blood pressure over 130/85 mmHg, fasting triglyceride (TG) level over 150 mg/dl, fasting high-density lipoprotein (HDL) cholesterol level less than 40 mg/dl (men) or 50 mg/dl (women) and fasting blood sugar over 100 mg/dl.
  Obesity was defined as a BMI of ≥ 25.0 kg/m2 . Patients with a BMI of 18.5-<23.0 were considered normal weight; for those with a BMI of 23.0-<25.0 were overweight. The patients with normal weight and those who were overweight were collapsed into the non-obesity group.
  so this group of patients are metabolically unhealthy ( have three or more of metabolic syndrome criteria) and non obese with BMI 18.5 - <25
  Interventions: Diagnostic Test: 24 hour urinary protein
- metabolically unhealthy obesity ( MUO ): According to the NCEP ATP III definition, metabolic syndrome is present if three or more of the following five criteria are met: waist circumference over 40 inches (men) or 35 inches (women), blood pressure over 130/85 mmHg, fasting triglyceride (TG) level over 150 mg/dl, fasting high-density lipoprotein (HDL) cholesterol level less than 40 mg/dl (men) or 50 mg/dl (women) and fasting blood sugar over 100 mg/dl.
  Obesity was defined as a BMI of ≥ 25.0 kg/m2 . Patients with a BMI of 18.5-<23.0 were considered normal weight; for those with a BMI of 23.0-<25.0 were overweight. The patients with normal weight and those who were overweight were collapsed into the non-obesity group.
  so this group of patients are metabolically unhealthy but they are obese with BMI of ≥ 25.0 kg/m2
  Interventions: Diagnostic Test: 24 hour urinary protein

INTERVENTIONS:
Diagnostic Test: 24 hour urinary protein — proteinuria and renal function impairment will be detected in patients of four groups
  Other Names: kidney function test : urea and creatinine; eGFR

SUMMARY:
1. Comparison between the 4 groups of metabolic phenotypes of obesity as regard the presence and frequency of DKD
2. Relation between DKD , obesity (BMI) and metabolic risk factors in patients with type 2 DM

DETAILED DESCRIPTION:
Diabetes is the major cause of chronic kidney disease in industrialized countries. Individuals with diabetes and CKD are at a higher risk of developing End Stage Renal Disease and experiencing cardiovascular death. Type 2 DM complications are predicted by low estimated glomerular filtration rate and high urine albumin excretion(1).

Diabetic kidney disease is the primary cause of kidney failure globally, affecting 25% to 40% of persons with diabetes mellitus . Early diagnosis of high-risk patients is crucial due to the high-risk of progressive deterioration of kidney function leading to end-stage kidney disease, which ultimately requires kidney replacement therapy (2).

DKD risk factors include non modifiable factors like age , gender , race , genetics and modifiable factors like obesity and lifestyle. Obesity is typically associated with metabolic diseases such as hyperglycemia, dyslipidemia, and high blood pressure. Obesity's impact on renal insufficiency is debated ,and may be influenced by other metabolic abnormalities(3).

Metabolic phenotypes of obesity based on the BMI-based categories (non-obesity, obesity) and metabolic status (metabolically healthy status or metabolically unhealthy status): metabolically Healthy non-obesity (MHNO), metabolically healthy obesity (MHO), metabolically unhealthy non-obesity (MUNO) and metabolically unhealthy obesity (MUO)(3).

There is a strong correlation between obesity and the onset and course of chronic kidney disease, according to a number of population-based studies. the investigators think there are still unsolved issues about the connection between obesity and CKD(4).

so the study is concerned about detection of the relation between metabolic phenotypes of obesity and Diabetic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic adult patients admitted at Assiut university hospital divided into 4 groups of metabolic phenotypes according to obesity and metabolic status .

Exclusion Criteria:

1. Age less than 18
2. type 1 diabetes
3. those with a BMI <18.5 kg/m2
4. co-existing non-diabetic renal disease
5. Pregnancy and patients with malignancy
6. Urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic adult patients admitted at Assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Conclusion of the relationship between metabolic phenotypes of obesity and Diabetic kidney disease in type 2 diabetes Mellitus patients | Baseline
  conclusion the relation between metabolic phenotypes of obesity and diabetic kidney disease in type 2 diabetes mellitus patients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bentata Y, Latrech H, Abouqal R. Does body mass index influence the decline of glomerular filtration rate in diabetic type 2 patients with diabetic nephropathy in a developing country? Ren Fail. 2014 Jul;36(6):838-46. doi: 10.3109/0886022X.2014.899472. Epub 2014 Mar 27. PMID 24673339
- [Background] Jung CY, Yoo TH. Pathophysiologic Mechanisms and Potential Biomarkers in Diabetic Kidney Disease. Diabetes Metab J. 2022 Mar;46(2):181-197. doi: 10.4093/dmj.2021.0329. Epub 2022 Mar 24. PMID 35385633
- [Background] Zhao L, Zou Y, Wu Y, Cai L, Zhao Y, Wang Y, Xiao X, Yang Q, Yang J, Ren H, Tong N, Liu F. Metabolic phenotypes and risk of end-stage kidney disease in patients with type 2 diabetes. Front Endocrinol (Lausanne). 2023 May 10;14:1103251. doi: 10.3389/fendo.2023.1103251. eCollection 2023. PMID 37234807
- [Background] Evangelista LS, Cho WK, Kim Y. Obesity and chronic kidney disease: A population-based study among South Koreans. PLoS One. 2018 Feb 28;13(2):e0193559. doi: 10.1371/journal.pone.0193559. eCollection 2018. PMID 29489920